CLINICAL TRIAL: NCT05625906
Title: The Effectiveness of a Multi-media Experiential Training Programme in Advance Care Planning for Nurses Working in Acute Care Settings
Brief Title: Advance Care Planning Training for Nurses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Carmen Chan Yip Wing-han, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2018.610
Record Dates: First submitted 2022-11-06; First posted 2022-11-23 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Advance Care Planning
Keywords: Advance Care Planning; acute care settings; experiential learning; nurse training programme

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): will receive a multi-media experiential training programme.
  Interventions: Other: Multi-media experiential training programme
- control group (No Intervention): will NOT receive a multi-media experiential training programme

INTERVENTIONS:
Other: Multi-media experiential training programme — 1. Webpage and mobile applications of training material on ACP, to be offered four weeks before the workshop
  2. A three-hour multimedia workshop (8-10 nurses per group) including enhanced lectures and a role play encounter with standardised patients. Immediate feedback on their quality of decision support skills will be given. The workshops will be delivered by an experienced advance practice nurse with a palliative care specialty.
  3. Writing a reflective journal after the role play with standardised patients
  Arms: Intervention group

SUMMARY:
The aims of this study are to examine the effectiveness of a multi-media experiential training programme in advance care planning (ACP) for nursing staff in acute care settings. The main questions it aims to answer are:

* can the programme enhance nurses' decision-support skills
* can the programme strengthen nurses' knowledge and confidence, and improve their attitude toward ACP?

Researchers will compare the participants in the intervention group (receive training programme) with those who are in the control group (receive no intervention) to evaluate the effectiveness of the programme.

DETAILED DESCRIPTION:
The study adopts a cluster randomised controlled trial with 12 weeks (T2) and 24 weeks (T3) follow-ups. A total of 234 eligible nurses working in 26 acute care hospital wards will be randomised at ward level in a 1:1 ratio into either control or intervention arms. Guided by the Theory of Planned Behaviour, we will conduct path analysis to assess the role of nurses' knowledge, attitudes and confidence on the nurses' skill performance on decision support after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* registered nurse with at least two years' clinical experience

Exclusion Criteria:

* had prior specialty training in Advance Care Planning communication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Nurse's decision support skills as assessed by the Brief Decision Support Analysis Tool (DSAT10) | Baseline
  DSAT10 instrument is an observational feedback tool for evaluating decisional support interactions between health care workers and patients. The DSAT-10 includes 16 items divided into five domains of: Decision-Making Status; Knowledge of Options, Risks, and Benefits; Values Associated with Outcomes of Options. Scores range from zero to ten, with higher scores indicating more decisional support being verbalized during the patient-provider interaction.
Nurse's decision support skills as assessed by the Brief Decision Support Analysis Tool (DSAT10) | immediate post-intervention
  DSAT10 instrument is an observational feedback tool for evaluating decisional support interactions between health care workers and patients. The DSAT-10 includes 16 items divided into five domains of: Decision-Making Status; Knowledge of Options, Risks, and Benefits; Values Associated with Outcomes of Options. Scores range from zero to ten, with higher scores indicating more decisional support being verbalized during the patient-provider interaction.

SECONDARY OUTCOMES:
Nurses' attitudes towards Advance Care Planning | Baseline
  Nurses' attitudes towards ACP will be measured by nine five-point Likert scale items with 1=strongly disagree and 5= strongly agree. Higher scores indicate a more positive attitude. The scale was developed and validated by Putman-Casdorph et al . The nine items cover topics such as the perceived helpfulness of ACP, and worries about the legal consequences of limiting treatment.
Nurses' attitudes towards Advance Care Planning | immediate post-intervention
  Nurses' attitudes towards ACP will be measured by nine five-point Likert scale items with 1=strongly disagree and 5= strongly agree. Higher scores indicate a more positive attitude. The scale was developed and validated by Putman-Casdorph et al . The nine items cover topics such as the perceived helpfulness of ACP, and worries about the legal consequences of limiting treatment.
Nurses' attitudes towards Advance Care Planning | 12 weeks post-intervention
  Nurses' attitudes towards ACP will be measured by nine five-point Likert scale items with 1=strongly disagree and 5= strongly agree. Higher scores indicate a more positive attitude. The scale was developed and validated by Putman-Casdorph et al . The nine items cover topics such as the perceived helpfulness of ACP, and worries about the legal consequences of limiting treatment.
Nurses' knowledge of Advance Care Planning | Baseline
  Knowledge of advance care planning and advance directives will be assessed by a 10-item true / false questionnaire which is developed taking reference with Siu et al. and Yee et al. The knowledge test will be validated by an expert panel including academics and clinicians.
Nurses' knowledge of Advance Care Planning | immediate post-intervention
  Knowledge of advance care planning and advance directives will be assessed by a 10-item true / false questionnaire which is developed taking reference with Siu et al. and Yee et al. The knowledge test will be validated by an expert panel including academics and clinicians.
Nurses' knowledge of Advance Care Planning | 12 weeks post-intervention
  Knowledge of advance care planning and advance directives will be assessed by a 10-item true / false questionnaire which is developed taking reference with Siu et al. and Yee et al. The knowledge test will be validated by an expert panel including academics and clinicians.
Nurses' knowledge of Advance Care Planning | 24 weeks post-intervention
  Knowledge of advance care planning and advance directives will be assessed by a 10-item true / false questionnaire which is developed taking reference with Siu et al. and Yee et al. The knowledge test will be validated by an expert panel including academics and clinicians.
Nurses' level of confidence to conduct Advance Care Planning | Baseline
  Nurses' level of confidence to conduct ACP will be measured by a single item five-point Likert scale with 1= not confident at all to 5 = extremely confident .
Nurses' level of confidence to conduct Advance Care Planning | immediate post-intervention
  Nurses' level of confidence to conduct ACP will be measured by a single item five-point Likert scale with 1= not confident at all to 5 = extremely confident .
Nurses' level of confidence to conduct Advance Care Planning | 12 weeks post-intervention
  Nurses' level of confidence to conduct ACP will be measured by a single item five-point Likert scale with 1= not confident at all to 5 = extremely confident .
Nurses' level of confidence to conduct Advance Care Planning | 24 weeks post-intervention
  Nurses' level of confidence to conduct ACP will be measured by a single item five-point Likert scale with 1= not confident at all to 5 = extremely confident .
Nurses' satisfaction with the training programme | immediate post intervention
  Nurses' satisfaction with the training programme will be assessed by an eight-item five-point Likert scale with 1=strongly disagree and 5= strongly agree at post-test only. Higher scores indicate higher satisfaction. The scale is developed with reference to So et al. and has been validated by an expert panel including academics and clinicians.
Actual experience of Advance Care Planning in the last 12 weeks | Baseline
  Actual experience in ACP discussion will be measured by this question: "How many times have you participated in ACP discussion with your patients in the last 12 weeks?" In addition, documentation of the ACP discussion in the last 12 weeks will be retrieved from patients' medical records.
Actual experience of Advance Care Planning in the last 12 weeks | 12 weeks post-intervention
  Actual experience in ACP discussion will be measured by this question: "How many times have you participated in ACP discussion with your patients in the last 12 weeks?" In addition, documentation of the ACP discussion in the last 12 weeks will be retrieved from patients' medical records.
Actual experience of Advance Care Planning in the last 12 weeks | 24 weeks post-intervention
  Actual experience in ACP discussion will be measured by this question: "How many times have you participated in ACP discussion with your patients in the last 12 weeks?" In addition, documentation of the ACP discussion in the last 12 weeks will be retrieved from patients' medical records.
Adherence to patients' expressed preference for care | 12 weeks post-intervention
  measured by this question: Please circle the following to describe health care professionals' adherence to patients' expressed preference for care :
Adherence to patients' expressed preference for care | 24 weeks post-intervention
  measured by this question: Please circle the following to describe health care professionals' adherence to patients' expressed preference for care :

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Chan Yip Wing-han, Principal Investigator — Chinese University of Hong Kong
Locations (8):
- Hong Kong (8):
  - United Christian Hospital, Kwun Tong
  - Queen Elizabeth Hospital, Mong Kok
  - Prince of Wales Hospital, Shatin
  - Shatin cheshire home, Shatin
  - Shatin Hospital, Shatin
  - Haven of Hope Hospital, Tseung Kwan O
  - Tuen Mun Hospital, Tuenmen
  - Grantham Hospital, Wong Chuk Hang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Putman-Casdorph H, Drenning C, Richards S, Messenger K. Advance directives: evaluation of nurses' knowledge, attitude, confidence, and experience. J Nurs Care Qual. 2009 Jul-Sep;24(3):250-6. doi: 10.1097/NCQ.0b013e318194fd69. PMID 19525766
- [Background] Siu MW, Cheung TY, Chiu MM, Kwok TY, Choi WL, Lo TK, Ting WM, Yu PH, Cheung CY, Wong JG, Shua SE. The preparedness of Hong Kong medical students towards advance directives and end-of-life issues. East Asian Arch Psychiatry. 2010 Dec;20(4):155-62. PMID 22348923
- [Background] So WKW, Kwong ANL, Chen JMT, Chan JCY, Law BMH, Sit JWH, Chan CWH. A Theory-Based and Culturally Aligned Training Program on Breast and Cervical Cancer Prevention for South Asian Community Health Workers: A Feasibility Study. Cancer Nurs. 2019 Mar/Apr;42(2):E20-E30. doi: 10.1097/NCC.0000000000000543. PMID 28945633